CLINICAL TRIAL: NCT02753673
Title: Patient Expectations of Breast Conserving Therapy: Broadening a Patient Reported Outcomes Instrument
Brief Title: Developing a New Questionnaire About Patient Expectations of Breast Conserving Therapy
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Hospital for Special Surgery, New York (Other); McMaster University (Other)
Responsible Party: Sponsor
Other Study IDs: 16-325
Record Dates: First submitted 2016-04-22; First posted 2016-04-28 (Estimated); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer
Keywords: Breast Conserving Therapy; Reported Outcomes Instrument; 16-325
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Breast Cancer: The assessments are all qualitative. The assessments include an in-person, open-ended qualitative interview, during which the interviewer will use an interview guide to ensure that all relevant topics are discussed. Participants will also complete the Patient Expectations with Breast Reconstruction questionnaire using the think-aloud technique in order to identify which questions reflect the expectations of BCT patients, which questions need modification to reflect the expectations of BCT patients and which questions are not appropriate for BCT patients. The responses to the expectations questionnaire for this portion of the interview will not be recorded or analyzed; only the participants' thoughts and opinions about the questions will be recorded.
  Interventions: Behavioral: qualitative interviews with patients; Behavioral: questionnaires

INTERVENTIONS:
Behavioral: qualitative interviews with patients
Behavioral: questionnaires

SUMMARY:
The purpose of this study is to develop a questionnaire to measure patient expectations of breast-conserving therapy (breast-conserving surgery and radiation). This questionnaire will assist both surgeons and patients by helping provide valuable information to patients about what to expect during and after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18-75
* Patients who are scheduled to undergo lumpectomy at MSKCC as part of breast conserving therapy for invasive breast cancer OR who have completed BCT (lumpectomy and radiation) at least 6 months prior to recruitment

Exclusion Criteria:

* Inability to speak or understand English
* Inability to provide meaningful informed consent due to physical, cognitive, or psychiatric disability
* Patients undergoing lumpectomy without radiation

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MSKCC clinics
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2016-04-20 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2020-04-13 (Actual)

PRIMARY OUTCOMES:
measure patient expectations of breast-conserving therapy | 1 year
  This study aims to develop the Patient Expectations with Breast-Conserving Therapy questionnaire. New questionnaire content will be generated using qualitative research methods. Interview data will be analyzed using a grounded theory approach, which involves generating codes, categories, and themes inductively, rather than imposing a priori assumptions or classifications on the data.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L Pusic, MD, MHS,FRCSC, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/